CLINICAL TRIAL: NCT06313164
Title: The Impact of Oral Glutathione on Oxidative Damage and Glycated Hemoglobin (HbA1c) Levels in Type 2 Diabetes Patients: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: The Impact of Oral Glutathione on Oxidative Damage and Glycated Hemoglobin (HbA1c) Levels in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW009
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: oxidative stress; glutathione; antioxidants; preventive supplementation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enhanced L-gluthathione group (Experimental)
  Interventions: Dietary Supplement: enhanced glutathione
- placebo group (Placebo Comparator)
  Interventions: Other: placebo comparator

INTERVENTIONS:
Dietary Supplement: enhanced glutathione — L-glutathione (in combination with tannin, low molecular weight chitosan and polyethylene glycol)
  Arms: enhanced L-gluthathione group
Other: placebo comparator — placebo group
  Arms: placebo group

SUMMARY:
This trial aims to assess the effectiveness of L-glutathione, supplemented with bioavailability boosters (tannin, low molecular weight chitosan, and polyethylene glycol), on improving antioxidant levels and glycemic control in patients with type 2 diabetes (T2D). The study is designed as a randomized, double-blind, placebo-controlled trial intending to enroll 240 T2D patients. The primary objective is to measure changes from baseline to 180 days in several key biomarkers, including endogenous reduced glutathione (GSH), oxidized glutathione (GSSG), 8-hydroxydeoxyguanosine (8-OHdG), and glycated hemoglobin (HbA1c), along with other metabolic parameters.

Hypothesis: The anticipated outcome is a significant increase in GSH levels and a decrease in markers of oxidative damage among participants receiving L-glutathione compared to those in the placebo group, potentially indicating improved antioxidant defenses and some effects on glycemic regulation in T2D patients. This trial aims to fill gaps in current research regarding the role of L-glutathione supplementation in managing oxidative stress and metabolic control in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* subjects with diabetes mellitus type 2 with confirmed levels of glycated hemoglobin (HbA1c) ≥ 6.5%

Exclusion Criteria:

* pregnancy and breastfeeding
* heavy smoking: Individuals consuming more than 20 cigarettes per day;
* excessive alcohol consumption: Participants who consume alcohol in excess of established limits, defined as more than 14 standart doses for men and 7 for woman;
* active clinical infections
* recent cardiovascular events: Individuals who suffered from cardiovascular event in the last 6 months;
* subjects receiving antioxidant drugs or dietary supplements;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Сhanged glutathione (GSH) levels in erythrocyte hemolysate change in patients with type 2 diabetes mellitus | 180 days

SECONDARY OUTCOMES:
Oxidized Glutathione (GSSG) Levels Change in Patients with Type 2 Diabetes Mellitus | 180 days
8-Oxoguanine (8-OHdG) Levels Change in Patients with Type 2 Diabetes Mellitus | 180 days
Glycated Hemoglobin Concentration (HbA1c) Change in Patients with Type 2 Diabetes Mellitus | 180 days
Fasting Glucose (FPG) Levels Change in Patients with Type 2 Diabetes Mellitus | 180 days
Postprandial Glucose (PPG) Levels Change in Patients with Type 2 Diabetes Mellitus | 180 days
Fasting Insulin (FPI) Levels Change in Patients with Type 2 Diabetes Mellitus | 180 days
Postprandial Insulin (PPI) Levels Change in Patients with Type 2 Diabetes Mellitus | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia